CLINICAL TRIAL: NCT02479828
Title: The Effect of Fascia Iliaca Compartment Block in Acute and Chronic Pain Management in Hip Fracture Patients
Brief Title: Fascia Iliaca Compartment Block in Acute and Chronic Pain Management in Hip Fracture Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Asklepieion Voulas General Hospital (Other Government)
Responsible Party: Principal Investigator, Maria Diakomi, Anesthesiologist, Asklepieion Voulas General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 7533
Record Dates: First submitted 2015-06-10; First posted 2015-06-24 (Estimated); Last update posted 2019-03-12 (Actual); Status verified 2019-03

CONDITIONS: Chronic Hip Pain
MeSH Terms: interventions — Ropivacaine; Ultrasonography

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fascia iliaca compartment block (FICB) (Active Comparator): Under ultrasound guidance performing fascia iliaca compartment block, in which 40 ml ropivacaine 0,5% are injected under the fascia iliaca.
  Interventions: Drug: Fascia iliaca compartment block; Drug: Ropivacaine; Device: ultrasound
- Placebo (not FICB) (Placebo Comparator): Half of the patients will not receive FICB
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fascia iliaca compartment block — 40 ml ropivacaine 0,5% injected under fascia iliaca using ultrasound
  Arms: Fascia iliaca compartment block (FICB)
Drug: Ropivacaine
  Arms: Fascia iliaca compartment block (FICB)
Device: ultrasound
  Arms: Fascia iliaca compartment block (FICB)
Drug: Placebo
  Arms: Placebo (not FICB)

SUMMARY:
This study evaluates the effect of fascia iliaca compartment block (FICB) in the management of acute post -surgical pain in hip fracture patients and in the appearance of chronic post -surgical hip pain, by means of von Korff Graded Chronic Pain Scale -modified for hip pain in Greek.

Half of the patients will not receive fascia iliaca compartment block.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-III (American Society of Anesthesiologists classification)
* intertrochanteric fractures
* fractures of femoral neck

Exclusion Criteria:

* existing pain in hip Joint to be operated
* cognitive or mental disorder
* administration of analgesic drugs prior surgery
* contraindications of spinal anesthesia
* refusal to participate in the study

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Acute postsurgical pain after hip fracture surgery | 48 hours
  Acute pain will be evaluated using the Numeric Rating Scale- NRS (0=no pain, 10= Extremely strong pain) at rest and in motion.
Chronic postsurgical pain after hip fracture surgery | 6 months
  3 and 6 months after surgery the patient or patient's relative will be asked on telephone to complete Von Korff Graded Chronic scale modified for hip pain

CONTACTS AND LOCATIONS:
Overall Officials: MARIA DIAKOMI, Principal Investigator — Asklepieion General Hospital
Locations (1):
- Asklepieion General Hospital, Athens, Voula, Greece

REFERENCES:
- [Derived] Guay J, Kopp S. Peripheral nerve blocks for hip fractures in adults. Cochrane Database Syst Rev. 2020 Nov 25;11(11):CD001159. doi: 10.1002/14651858.CD001159.pub3. PMID 33238043